CLINICAL TRIAL: NCT06022978
Title: Submucosal Saline Injection Followed by Endoscopic Ultrasound Versus Endoscopic Ultrasound Only for Distinguishing Between T1a and T1b Esophageal Cancer
Brief Title: Submucosal Saline Injection Followed by Endoscopic Ultrasound
Acronym: EUS-SSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Zhejiang Cancer Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); Shandong Cancer Hospital and Institute (Other); Xinqiao Hospital of Chongqing (Other); Sir Run Run Shaw Hospital (Other); The Second Affiliated Hospital of Shaanxi University of Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Jian-jun Li, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FXY-068
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Esophageal Cancer
Keywords: Submucosal Saline Injection; Endoscopic Ultrasound; Early Esophageal Cancer; Staging
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EUS only (No Intervention): The enrolled patients will accept ordinary EUS only.
- EUS+SSI (Experimental): The enrolled patients will be accepted submucosal injection of saline（SSI）,then EUS will be performed.
  Interventions: Procedure: Submucosal Saline Injection
- BLI+ME/EUS+SSI (Experimental): The enrolled patients will be accepted ordinary endoscope using blue laser Imaging and magnified ensocope system(BLI+ME), firstly. If B3 type intra pillary capillary loops (IPCL) was observed, then the procedure would be finished (no EUS or EUS+SSI) . If B1 or B2 type IPCL was observed, then EUS+SSI would be performed.
  Interventions: Procedure: Submucosal Saline Injection; Procedure: Blue laser Imaging and Magnifying Endoscopy

INTERVENTIONS:
Procedure: Submucosal Saline Injection — Inject 3-5 mL of saline into the submucosa within 10 minutes using a single-use 22G mucosal needle. The puncture point is located 0.5 cm from the edgeof the lesion, and the saline injection is stopped when the esophageal mucosa is elevated by approximately 1 cm.
  Arms: BLI+ME/EUS+SSI; EUS+SSI
Procedure: Blue laser Imaging and Magnifying Endoscopy — It is a new system for image-enhanced endoscopy using laser light. By clicking a button on the endoscope only , endoscopists can electronically stain and magnify the digestive tract lesions. This system can help endoscopists observe leisons more clearly and improve diagnosic accuracy.
  Arms: BLI+ME/EUS+SSI

SUMMARY:
Endoscopic ultrasound (EUS) is unsatisfactory in distinguishing between T1a and T1b stage esophageal squamous cell carcinoma (ESCC). Consequently, the National Comprehensive Cancer Network guidelines recommend endoscopic resection (ER) as a diagnostic tool for substaging T1 stage ESCC. However, as an invasive approach, diagnostic ER is not an optimal approach especially for T1b cases as most of them might not be fully cured by ER. It is necessary to develop reliable and less invasive methods to distinguish between T1a and T1b stage ESCC. In our previous unicentral trial, we found that submucosal saline injection (SSI) significantly improved the diagnostic accuracy of EUS in differentiating between T1a and T1b stage ESCC. It can be used as an alternative to diagnostic ER for preoperative substaging T1 stage ESCC cases in remote regions where few endoscopists are able to perform diagnostic ER. The use of EUS and SSI would help T1b stage patients avoid invasive diagnostic ER.

Therefore, we aim to conduct a multi-center clinical trail to examine whether SSI can improve traditional EUS accuracy in distinguishing between T1a and T1b stage ESCC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old, no gender limited;
* Patients with esophageal squamous cell carcinoma who be confirmed by ordinary endoscopy and pathologic biopsy;
* Patients who agree to accept endoscopic resection or surgical excision of the lesion in esophagus;
* patients with normal cardio-pulmonary function and normal coagulative function,are predicted to be tolerated anesthesia and surgery;
* patients who understand test purpose, volunteer to join these study and sign the consent inform.

Exclusion Criteria:

* Patients with stages of T2, T3, or T4 displayed by EUS;
* Patients who can't tolerate endoscopy and surgical treatment for various reasons;
* Patients who have distant metastasis, or multiple source of malignant tumors;
* Patients with blood coagulative disorder;
* Patients don't accept the endoscopic examination or surgical treatment;
* Patients with poor compliancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy for T1a and T1b staging | Participants will be followed for the duration of hospital stay in order to accept endosopic or surgical resection , an expected average of 10 days
  The stages judged from EUS or EUS+SSI or BLI+ME/EUS+SSI will be compared with the pathological results after endoscopic or surgical resection. So the sensitivity, specificity, positive predictive value, negative predictive value and diagnostic accuracy of the three groups for early esophageal cancer will be measured respectivly.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-jun Li, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol